CLINICAL TRIAL: NCT04160494
Title: A Phase 1 Trial of D2C7-IT in Combination With Atezolizumab in Recurrent WHO Grade IV Malignant Glioma
Brief Title: D2C7-IT With Atezolizumab for Recurrent Gliomas
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Darell Bigner (Other)
Collaborators: Istari Oncology, Inc. (Industry); National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Darell Bigner, E. L. and Lucille F. Jones Cancer Distinguished Research Professor, in the School of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00101898; FOR0003 (Other: National Cancer Institute)
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Malignant Glioma
Keywords: D2C7; D2C7-IT; Atezolizumab; Randazzo; Glioblastoma; Glioma; Bigner; Pro00101898; Genentech; CTEP; Duke; Landi
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — D2C7-(scdsFv)-PE38KDEL; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- D2C7-IT (6920 ng/mL) + Atezolizumab (Experimental): Single D2C7-IT convection-enhanced delivery (CED) infusion (6920 ng/mL) plus atezolizumab (1200 mg) intravenous (IV) infusions every three weeks for up to two years
  Interventions: Drug: D2C7-IT (6920 ng/mL via convection-enhanced delivery); Drug: Atezolizumab (1200 mg every three weeks)
- D2C7-IT (4613.2 ng/mL) + Atezolizumab (Experimental): Single D2C7-IT convection-enhanced delivery (CED) infusion (4613.2 ng/mL) plus atezolizumab (1200 mg) intravenous (IV) infusions every three weeks for up to two years
  Interventions: Drug: Atezolizumab (1200 mg every three weeks); Drug: D2C7-IT (4613.2 ng/mL via convection-enhanced delivery)

INTERVENTIONS:
Drug: D2C7-IT (6920 ng/mL via convection-enhanced delivery) — dual-specific mAB
  Arms: D2C7-IT (6920 ng/mL) + Atezolizumab
Drug: Atezolizumab (1200 mg every three weeks) — programmed cell death ligand 1 (PD-L1) blocking antibody
  Other Names: Tecentriq
Drug: D2C7-IT (4613.2 ng/mL via convection-enhanced delivery) — dual-specific mAB
  Arms: D2C7-IT (4613.2 ng/mL) + Atezolizumab

SUMMARY:
This is a phase 1 study of atezolizumab in combination with D2C7-IT, a dual-specific monoclonal antibody (mAB) with a high affinity for both EGFRwt- and EGFRvIII-expressing cells, in patients with recurrent World Health Organization (WHO) grade IV malignant glioma at the Preston Robert Tisch Brain Tumor Center (PRTBTC) at Duke.

DETAILED DESCRIPTION:
Approximately eighteen patients with recurrent WHO grade IV malignant glioma will receive atezolizumab and D2C7-IT to determine the impact of the combination of D2C7-IT and atezolizumab on safety. D2C7-IT will be delivered intratumorally by Convection Enhanced Delivery (CED) using an intracerebral catheter placed within the enhancing portion of the tumor. The dose of D2C7-IT was reduced from 6920 ng/mL to 4613.2 ng/mL after the first 4 patients as a precaution due to safety events experienced by these 4 patients.

Atezolizumab will be administered according to the FDA-approved dosing schedule of 1200 mg intravenously every 3 weeks, beginning ~2 weeks after the D2C7-IT infusion.

Toxicity will be carefully monitored for each patient while they are on study for at least a year after D2C7-IT treatment or for at least 30 days after the final dose of atezolizumab if the patient continues atezolizumab on-study for longer than a year post-D2C7-IT. Of particular interest will be the incidence of adverse events that occur during the first 28 days after D2C7-IT treatment and the inflammatory events that occur during the first year after D2C7-IT treatment.

The most common risks associated with D2C7-IT are effects related to tumor necrosis, neurologic changes (including changes in function, new or increased seizures, swelling of the brain, and injury to blood vessels), effects related to catheter placement or removal, and effects related to fluid infusion into the brain. The most common risks associated with atezolizumab are fatigue, decreased appetite, diarrhea, and nausea. Because atezolizumab works with the immune system, it can cause the immune system to attack normal organs or tissue and affect how they work.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a recurrent supratentorial WHO grade IV malignant glioma based on imaging studies
* Prior histopathology confirmed recurrent supratentorial WHO grade IV malignant glioma
* Patient or partner(s) meets one of the following criteria:

  1. Non-childbearing potential (i.e. not sexually active, physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile, or any male who has had a vasectomy). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal l ligation. Postmenopausal for purposes of this study is defined as 1 year without menses; or,
  2. Childbearing potential and agrees to use one of the following methods of birth control: approved hormonal contraceptives that do not contain estrogen (e.g., birth control pills, patches, implants, or infusions), an intrauterine device, or a barrier method of contraception (e.g., a condom or diaphragm) used with spermicide.
* Age ≥ 18 years of age at the time of entry into the study
* Karnofsky Performance Score (KPS) ≥ 70%
* Hemoglobin ≥ 9 g/dl prior to biopsy
* Platelet count ≥ 100,000/µl unsupported is necessary for eligibility on the study; however, because of risks of intracranial hemorrhage with catheter placement, platelet count ≥ 125,000/µl is required for the patient to undergo biopsy and catheter insertion, which can be attained with the help of platelet transfusion
* Neutrophil count ≥ 1000 cells/mm3 prior to biopsy
* Creatinine ≤ 1.5 x upper limit of normal (ULN) range prior to biopsy
* Total bilirubin ≤ 1.5 x ULN prior to biopsy, s (Exception: Patient has known Gilbert's Syndrome or patient has suspected Gilbert's Syndrome, for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3.0 x ULN is acceptable.)
* AST (aspartate aminotransferase)/ALT (alanine aminotransferase) ≤ 2.5 x ULN prior to biopsy
* Prothrombin and Partial Thromboplastin Times ≤ 1.2 x ULN prior to biopsy. Patients with prior history of thrombosis/embolism are allowed to be on anticoagulation, understanding that anticoagulation will be held in the perioperative period per the neurosurgical team's recommendations. Low molecular weight heparin (LMWH) is preferred. If a patient is on warfarin, the international normalized ratio (INR) is to be obtained and value should be below 2.0 prior to biopsy.
* At the time of biopsy, prior to administration of D2C7-IT, the presence of recurrent tumor must be confirmed by histopathological analysis
* A signed informed consent form approved by the Institutional Review Board (IRB) will be required for patient enrollment into the study. Patients must be able to read and understand the informed consent document and must sign the informed consent indicating that they are aware of the investigational nature of this study
* Able to undergo brain MRI with and without contrast

Exclusion Criteria:

* Females who are pregnant or breast-feeding
* Patients with an impending, life-threatening cerebral herniation syndrome, based on the assessment of the study neurosurgeons or their designate
* Patients with severe, active co-morbidity, defined as follow:

  1. Patients with an active infection requiring intravenous treatment or having an unexplained febrile illness (Tmax > 99.5°F/37.5°C)
  2. Patients with known immunosuppressive disease or known human immunodeficiency virus infection
  3. Patients with unstable or severe intercurrent medical conditions such as severe heart disease (New York Heart Association Class 3 or 4)
  4. Patients with known lung (forced expiratory volume in the first second of expiration (FEV1) < 50%) disease or uncontrolled diabetes mellitus
  5. Patients with albumin allergy
  6. Patients with severe (i.e., anaphylactic) gadolinium allergy. Patients with mild allergies (e.g., rash only) will be pretreated with acetaminophen and diphenhydramine prior to injection of the contrast agent
* Patients may not have received chemotherapy or bevacizumab ≤ 4 weeks [except for nitrosourea (6 weeks) or metronomic dosed chemotherapy such as daily etoposide or cyclophosphamide (1 week)] prior to starting the study drug unless patients have recovered from side effects of such therapy. Patients should discontinue use of tumor- treating fields (TTFs), such as Optune™, at least one week prior to D2C7-IT infusion.
* Patients may not have received immunotherapy ≤ 4 weeks prior to starting the study drug unless patients have recovered from side effects of such therapy
* Patients may not be less than 12 weeks from radiation therapy, unless progressive disease outside of the radiation field or 2 progressive scans at least 4 weeks apart or histopathologic confirmation
* Patients who have not completed all standard of care treatments, including surgical procedure and radiation therapy (at least 59 Gy)

  1. If the MGMT promoter in their tumor is known to be unmethylated, patients are not mandated to have received chemotherapy prior to participating in this trial
  2. If the MGMT promoter in their tumor is known to be methylated or the MGMT promoter methylation status is unknown at time of screening, patients must have received at least one chemotherapy regimen prior to participating in this trial
* Patients with neoplastic lesions in the brainstem, cerebellum, or spinal cord; radiological evidence of active (growing) disease (active multifocal disease); extensive subependymal disease (tumor touching subependymal space is allowed); tumor crossing the midline or leptomeningeal disease
* Patients on greater than 4 mg per day of dexamethasone within the 2 weeks prior to the D2C7-IT infusion
* Patients with worsening steroid myopathy (history of gradual progression of bilateral proximal muscle weakness, and atrophy of proximal muscle groups)
* Patients with prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
* Patients with a known history of hypersensitivity to atezolizumab, or any components of atezolizumab
* Patients with active autoimmune disease requiring systemic immunomodulatory treatment within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with an unacceptable adverse event | 2 years
  An unacceptable adverse event includes any Grade 3 or any Grade 4 toxicity that is not reversible within 2 weeks, any life-threatening event, or any treatment-related death. Also included are any grade 2 or higher serious autoimmune toxicities, particularly those affecting vital organs (e.g. cardiac, renal, CNS) if it occurs within 2 weeks of any protocol treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Landi, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center — https://tischbraintumorcenter.duke.edu/
- See also: Duke Health — https://www.dukehealth.org/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT04160494/ICF_000.pdf